CLINICAL TRIAL: NCT01436864
Title: A Phase 3 Clinical Trial of Intravitreal Injections of Human Recombinant Vascular Endothelial Growth Factor Receptor-Fc Fusion Protein in Patients With Choroidal Neovascularization Secondary to Age-related Macular Degeneration
Brief Title: A Randomized, Double-masked, Multicenter,Sham-controlled, Safety and Efficacy Study of KH902 in Patients With Wet AMD
Acronym: PHOENIX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chengdu Kanghong Biotech Co., Ltd. (Industry)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KHSWKH902005
Record Dates: First submitted 2011-09-19; First posted 2011-09-20 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: Recombinant Human VEGF Receptor-Fc Fusion Protein (KH902); age-related macular degeneration (AMD); choroidal neovascularization (CNV); intravitreal injection; best corrected visual acuity (BCVA); central retinal thickness
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 0.5 mg KH902 (Experimental): Patients will receive intravitreal injection of KH902 0.5mg/eye once per month for three times in the study eye, and then patients will receive 2 sham injections monthly, respectively, at the end of month 3 (visit 5), and following these injections you will receive intravitreal injection of KH902 once every three months, till month 12 (respectively at month 5, month 8 and month 11)
  Interventions: Biological: Recombinant Human VEGF Receptor-Fc Fusion Protein
- Sham-injection (Sham Comparator): Patients will receive sham injection once per month for three times, and then you will receive intravitreal injection of KH902 0.5mg/eye once per month for three times in the study eye, after three months' treatment they will receive intravitreal injection of KH902 once every three months, till month 12 (respectively at month 8 and month 11.
  Interventions: Biological: Recombinant Human VEGF Receptor-Fc Fusion Protein

INTERVENTIONS:
Biological: Recombinant Human VEGF Receptor-Fc Fusion Protein — Intravitreal injection of KH902 once per month

SUMMARY:
This study is designed to prove and confirm the efficacy and safety of multiple injections of human recombinant vascular endothelial growth factor receptor-Fc fusion protein (KH902) in patients with choroidal neovascularization due to neovascular age-related macular degeneration by comparing intravitreal injections of KH902 with sham-injections.

DETAILED DESCRIPTION:
AMD is the leading cause of severe vision loss in people over the age of 65 in the United States and other western countries. A quantity of documents indicate that neovascularization promoted by VEGF is the main cause of visual acuity decline. Patients are starving for a new drug which can notably improve VA with less administration frequency and lower treatment cost.

The new drug Recombinant Human VEGF Receptor-Fc Fusion Protein (KH902) is a gene fusion protein. The pre-clinical researches and phase II study showed that KH902 is well-tolerated,and safe, it is effective in inhibiting the growth, migration, pullulation of vascular endothelial cells and neovascularization induced by VEGF.

This study is designed to prove and confirm the efficacy and safety of multiple injections of KH902 in patients with choroidal neovascularization due to neovascular age-related macular degeneration by comparing intravitreal injections of KH902 with sham-injections.

ELIGIBILITY:
Inclusion Criteria:

* Signed the Informed Consent Form;
* Age ≥ 50 years of either gender;
* Total lesion size ≤ 30 mm2 of the study eye;
* BCVA score of the study eye between 73 and 19 letters;
* Clear ocular media and adequate pupil dilation to permit good quality fundus photographic imaging.
* BCVA score of the fellow eye ≥ 19 letters.

Exclusion Criteria:

* Current or previous non-exudative AMD diseases which affect the inspection and measurement of macular or the central visual acuity;
* Subretinal hemorrhage area≥ 50% of total lesion size;
* Scar or fibrosis area in study eyes ≥ 50% of total lesion size; or central foveal scar、fibrosis or atrophy of macular in the study eye;
* Presence of retinal pigment epithelial tear, retinal macular tractional, macular epiretinal membrane, and diagnosed with polypoidal choroidal vasculopathy in the study eye;
* Previous anti-VEGF drug treatment in the study eye within six months preceding screening; or anti-VEGF treatment in the fellow eye within three months before screening;
* Previous intraocular or periocular operations, excluding operations on eyelid without hampering the intravitreal injection in the study eye;
* Previous ophthalmologic operations in the study eye;
* Current active inflammation or infection in either eye;
* Uncontrolled previous or current glaucoma in either eye, or previous glaucoma filtering operation in the study eye;
* Current systemic administrations which may lead to toxicity in the crystalline lens;
* History of allergy or current allergic response;
* History of surgery within one month preceding enrollment;
* Infectious diseases need systemic administration;
* Systemic autoimmune diseases;
* Any uncontrolled clinical disorders;
* Patients of child-bearing potential do not adopted adequate contraception methods;
* Pregnant or nursing women;
* Patients should be excluded in the opinion of investigators;

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2011-08; Primary Completion 2012-12 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in BCVA | at month 3
  To evaluate the mean change from baseline in best-corrected visual acuity (BCVA) in KH902 treatment group and sham treatment group at month 3 and compare the difference between the values

SECONDARY OUTCOMES:
The incidence rate of adverse event | at month 3
  To evaluate the difference in safety assessment between Conbercept (KH902) group and Sham group at month 3.
Mean change of retinal thickness from baseline | at month 3
  To evaluate the mean change of retinal thickness from baseline in KH902 treatment group or sham treatment group at month 3.

CONTACTS AND LOCATIONS:
Overall Officials: Xun Xu, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (11):
- China (11):
  - First Affiliated Hospital of Fujian Medical College, Fuzhou, Fujian
  - Joint Shantou International Eye Center of Shantou University and The Chinese University of Hong Kong, Shantou, Guangdong
  - People's Hospital of Wuhan University, Wuhan, Hubei
  - Wuhan General Hospital of Guangzhou Military Command, Wuhan, Hubei
  - Wuxi Second People's Hospital, Wuxi, Jiangsu
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Ophthalmologic Hospital of Qingdao, Qingdao, Shandong
  - Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Affiliated Hospital of Wenzhou Medical College, Wenzhou, Zhejiang
  - Daping Hospital of the Third Military Medical University, Chongqing
  - Shanghai First People's Hospital, Shanghai